CLINICAL TRIAL: NCT05323591
Title: A Prospective, Non-interventional Study in Patients With Moderate to Severe Active Rheumatoid Arthritis in France Receiving Filgotinib for 2 Years
Brief Title: Prospective Observational Study of Filgotinib in Participants With Rheumatoid Arthritis in France
Acronym: PARROTFISH
Status: Active, not recruiting | Type: Observational
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: GLPG0634-CL-424; 49028 (Other: HMA-EMA Catalogues)
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: filgotinib; safety; effectiveness; patient-reported outcome
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Filgotinib: Participants will receive treatment for moderate to severe active RA with at least one dose of filgotinib in accordance with the product label.
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablets are administered in accordance with the product label
  Other Names: Jyseleca

SUMMARY:
An observational study to describe the effectiveness, safety, and patient-reported outcomes (PROs) in participants with moderate to severe active rheumatoid arthritis (RA) in France receiving filgotinib in real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 years with a diagnosis of moderate to severe active RA being prescribed filgotinib in accordance with the local treatment practices and product label for the first time.
* Female participants of childbearing potential must agree to use contraception while taking filgotinib as per product label.
* Participants must be willing and able to use an electronic device to complete the study PROs.
* Participant must sign and date the Informed Consent Form (ICF) before enrollment into the study.

Exclusion Criteria:

* Participation in any interventional or non-interventional study without prior approval from the Medical Lead. This does not preclude inclusion of participants enrolled to national registries.
* Female participant is pregnant or intending to become pregnant while taking filgotinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants aged ≥ 18 years with moderate to severe active RA receiving filgotinib who will be enrolled in France.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Treatment Persistence Rate | Month 24
  Treatment persistence rate at 24 months, defined as the percentage of participants continuing to receive filgotinib for 24 months from treatment initiation.

SECONDARY OUTCOMES:
Disease Activity: Percentage of Participants Achieving Disease Activity Score for 28 Joint Count Using C-Reactive Protein (DAS28[CRP]) ≤3.2 and/or Clinical Disease Activity Index (CDAI) ≤10 | Up to 24 months
Disease Activity: Percentage of Participants Achieving DAS28(CRP) ≤2.6 and/or CDAI ≤2.8 | Up to 24 months
Number of Participants With Adverse Events and Serious Adverse Events | Up to 24 months
Participants' Assessment of Pain: Pain Visual Analogue Scale (VAS) Score | Up to 24 months
Participants' Assessment of Fatigue: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score | Up to 24 months
Participants' Assessment of Work Activities Impairment: Work Productivity and Activity Impairment: Rheumatoid Arthritis (WPAI-RA) Score | Up to 24 months
Participants' Assessment of Rheumatoid Arthritis Impact of Disease (RAID) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfasigma Study Director, Study Director — Alfasigma S.p.A.
Locations (17):
- France (17):
  - CHU Amiens Picardie site Nord, Amiens
  - CHU de Amiens Picardie, Amiens
  - Hopital Avicenne AP-HP, Bobigny
  - CHU Bordeaux, Bordeaux
  - CH de Cahors, Cahors
  - Clinique de l'Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Hopital Sud Francilien Corbeil Essonne, Corbeil-Essonnes
  - Hopital Roger Salengro, Lille
  - CHU de Nice, Nice
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Hopital Saint Antoine, Paris
  - Hopital Cochin Service A, Paris
  - Hopital Robert Debre, Reims
  - CHU de Rouen, Rouen
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No